CLINICAL TRIAL: NCT07319715
Title: Combined Cervical Cerclage and Vaginal Progesterone May Readjust the Deregulated Cervicovaginal Fluid Inflammatory Milieu and Improve Outcomes of Twin Pregnant Women
Brief Title: Cerclage and Progesterone for Twin Pregnancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Adel Farag Al Kholy, Professor of Medical Biochemistry, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Rc 4.12.2022
Record Dates: First submitted 2025-12-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Twin Pregnancy With Antenatal Problem

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cervical Cerclage (CC) (Active Comparator): Participants in this arm undergo a McDonald cerclage technique. This involves placing a purse-string suture (No. 1 or 2 braided or monofilament) around the cervix to close the internal os. The suture is typically removed at 37 weeks of gestation.
  Interventions: Procedure: McDonald Cervical Cerclage
- Vaginal Progesterone Therapy (VPT) (Active Comparator): Participants receive 100 mg vaginal progesterone inserts (e.g., Endometrin) administered twice daily. This treatment continues until spontaneous labor occurs or until the 37th week of pregnancy.
  Interventions: Drug: Vaginal Progesterone Therapy (VPT)
- Combined Therapy (CC/VPT) (Active Comparator): Participants receive both the surgical Cervical Cerclage procedure and the daily Vaginal Progesterone inserts as described in the individual arms above.
  Interventions: Procedure: McDonald Cervical Cerclage; Drug: Vaginal Progesterone Therapy (VPT)

INTERVENTIONS:
Procedure: McDonald Cervical Cerclage — The procedure involves exposing the cervix and grasping it with ring forceps. A purse-string suture using No. 1 or 2 braided or monofilament material is placed at the 12 o'clock position with a curved needle. The needle is inserted at the junction of the vaginal epithelium and the cervix, approximately 2 cm above the external os and distal to the vesicocervical reflection. After 5-6 cautious bites, the stitch is pulled tight to close the internal os. The suture is typically removed at 37 weeks of gestation, provided there is no labor or membrane rupture.
  Arms: Cervical Cerclage (CC); Combined Therapy (CC/VPT)
Drug: Vaginal Progesterone Therapy (VPT) — Participants receive 100 mg vaginal progesterone inserts.
  Dosage & Frequency: One 100 mg insert administered twice daily.
  Duration: The treatment continues until the onset of spontaneous labor or until the 37th week of pregnancy.
  Arms: Combined Therapy (CC/VPT); Vaginal Progesterone Therapy (VPT)

SUMMARY:
Twin pregnancies face a high risk of complications, most notably preterm birth (delivery before 37 weeks), which is a major cause of infant death and illness globally. For women carrying twins who are identified as having a short cervical length (cervix measuring 25 millimeters or less), there is currently no single, highly effective preventative treatment. This study is a randomized clinical trial designed to determine if a combined therapy of Cervical Cerclage (a surgical stitch to support the cervix) and Vaginal Progesterone (a hormone medication) is more effective than standard care in preventing preterm birth and improving the overall health outcomes for both the mother and the babies. The trial will also investigate the biological basis of this effect by measuring specific inflammation markers (cytokines like Interleukin-1$\beta$, 6, 8, and Tumor Necrosis Factor-α) in the cervical fluid before and after the intervention, to see if the combined treatment helps to reduce harmful local inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Type of Pregnancy: Women with confirmed twin pregnancy (TP).
* Cervical Length: Short cervical length (CL) defined as ≤25 mm.
* Timing of Diagnosis: Short cervix detected via transvaginal ultrasound (TVU) at 11-13 weeks + 6 days, or detected during bi-weekly follow-up exams until 23 weeks + 6 days.
* Consent: Participants willing to undergo randomization and comply with the follow-up protocol.

Exclusion Criteria:

* Multiple Gestation (High Order): Triplet or higher-order pregnancies.
* Fetal/Uterine Complications: Polyhydramnios, premature rupture of membranes (PPROM), or known uterine abnormalities.
* Acute Symptoms: Vaginal bleeding, fever, or signs of fetal distress.
* Maternal Comorbidities: Pre-existing or gestational hypertension, and diabetes mellitus.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 59 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2025-06-14 (Actual)

PRIMARY OUTCOMES:
Success Rate of Treatment Regimens in Preventing Preterm Birth and/or Improving Pregnancy Duration | 6-7 Months
  The proportion of patients who achieved a pregnancy duration of 37 weeks or more and/or significantly delayed delivery, reflecting the effectiveness of the administered treatment regimens (Cervical Cerclage, Vaginal Progesterone, or Combined Therapy) in high-risk twin pregnancies.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Benha University, Banhā, Qalyubia Governorate, Egypt